CLINICAL TRIAL: NCT01242527
Title: Efficacy and Safety of Epanova® (Omefas) in Severe Hypertriglyceridemia
Brief Title: Epanova® for Lowering Very High Triglycerides
Acronym: EVOLVE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OM-EPA-003
Record Dates: First submitted 2010-11-15; First posted 2010-11-17 (Estimated); Results first posted 2013-09-06 (Estimated); Last update posted 2016-08-04 (Estimated); Status verified 2016-06

CONDITIONS: Severe Hypertriglyceridemia
Keywords: dyslipidemia; hyperlipidemia; omega-3 carboxylic acid
MeSH Terms: conditions — Hypertriglyceridemia; Dyslipidemias; Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- Epanova 2 g (Experimental)
  Interventions: Drug: omefas
- Epanova 3 g (Experimental)
  Interventions: Drug: omefas
- Epanova 4 g (Experimental)
  Interventions: Drug: omefas

INTERVENTIONS:
Drug: placebo — 4 capsules (1g) daily for 12 weeks
  Arms: placebo
Drug: omefas — 2 capsules (1g) + 2 placebo daily for 12 weeks
  Arms: Epanova 2 g
Drug: omefas — 3 capsules (1g) + 1 placebo daily for 12 weeks
  Arms: Epanova 3 g
Drug: omefas — 4 capsules (1g)daily for 12 weeks
  Arms: Epanova 4 g

SUMMARY:
The primary objective of the study is to determine the efficacy of Epanova (omefas) compared to placebo in lowering serum triglycerides in subjects with severe hypertriglyceridemia.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, >=18 years of age.
* Very high serum TG values in the range >=500 mg/dL and <2000 mg/dL (>=5.65 mmol/L and <22.60 mmol/L)

Exclusion Criteria:

* Allergy or intolerance to omega-3 fatty acids, omega-3-acid ethyl esters, or fish.
* Known lipoprotein lipase impairment or deficiency or apolipoprotein C-II deficiency or familial dysbetalipoproteinemia.
* Unable to discontinue use of omega-3 drugs/supplements.
* Unable to discontinue use of bile acid sequestrants, fibrates or niacin (other than niacin-containing vitamins <200 mg), or any supplement used to alter lipid metabolism.
* Women who are pregnant, lactating, or planning to become pregnant. Women of childbearing potential who are not using acceptable contraceptive methods.
* Use of tamoxifen, estrogens or progestins that has not been stable for >4 weeks prior to Visit 1.
* Use of oral or injected corticosteroids or anabolic steroids.
* History of pancreatitis.
* History of symptomatic gallstone disease, unless treated with cholecystectomy.
* Uncontrolled diabetes.
* Uncontrolled hypothyroidism or thyroid stimulating hormone (TSH).
* History of cancer (other than basal cell carcinoma) in the past 2 years.
* Cardiovascular event (i.e., myocardial infarction, acute coronary syndrome, new onset angina, stroke, transient ischemic attack, unstable congestive heart failure requiring a change in treatment) or revascularization procedure within six months prior to Visit 1.
* Use of anticoagulants (e.g. warfarin [Coumadin®], coumarin, heparin, enoxaparin, clopidogrel).
* Presence of an aortic aneurysm or resection of an aortic aneurysm within six months prior to Visit 1.
* Recent history (within six months prior to Visit 1) or current significant nephrotic syndrome, pulmonary, hepatic, biliary, gastrointestinal or immunologic disease.
* Poorly controlled hypertension.
* Any of the following laboratory criteria: serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST), glucose, glomerular filtration rate (GFR), platelet count,or hemoglobin outside of study range.
* Recent history (past 12 months) of drug abuse or alcohol abuse.
* Exposure to any investigational product, within 4 weeks prior to Visit 1.
* Presence of any other condition the Investigator believes would interfere with the subject's ability to provide informed consent, comply with study instructions, or which might confound the interpretation of the study results or put the subject at undue risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Davidson, MD, FACC, Study Director — Omthera Pharmaceuticals, Inc
Locations (56):
- United States (28):
  - National City, California
  - Sacramento, California
  - Manchester, Connecticut
  - Coral Gables, Florida
  - Hialeah, Florida
  - Miami, Florida
  - Ocala, Florida
  - St. Petersburg, Florida
  - Summerfield, Florida
  - Atlanta, Georgia
  - Addison, Illinois
  - Chicago, Illinois
  - Louisville, Kentucky
  - Auburn, Maine
  - Olive Branch, Mississippi
  - High Point, North Carolina
  - Salisbury, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Bristol, Tennessee
  - Johnson City, Tennessee
  - Kingsport, Tennessee
  - San Antonio, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
  - Olympia, Washington
- Denmark (4):
  - Copenhagen
  - Gentofte Municipality
  - Herlev
  - Viborg
- Hungary (6):
  - Baja
  - Budapest
  - Debrecen
  - Sátoraljaújhely
  - Székesfehérvár
  - Szikszó
- India (8):
  - Karnāl, Haryana
  - Bangalore, Karnataka
  - Banswada, Karnataka
  - Indore, Madhya Pradesh
  - Pune, Maharashtra
  - Jaipur, Rajasthan
  - Chennai, Tamil Nadu
  - Surat
- Netherlands (4):
  - Amsterdam
  - Groningen
  - Rotterdam
  - Utrecht
- Russia (3):
  - Moscow
  - Novosibirsk
  - Saint Petersburg
- Ukraine (3):
  - Kharkiv
  - Kiev
  - Zaporizhzhya

REFERENCES:
- [Derived] Kastelein JJ, Maki KC, Susekov A, Ezhov M, Nordestgaard BG, Machielse BN, Kling D, Davidson MH. Omega-3 free fatty acids for the treatment of severe hypertriglyceridemia: the EpanoVa fOr Lowering Very high triglyceridEs (EVOLVE) trial. J Clin Lipidol. 2014 Jan-Feb;8(1):94-106. doi: 10.1016/j.jacl.2013.10.003. Epub 2013 Oct 14. PMID 24528690

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period started April 2011 and the last subject visit was February 2012. All subjects were qualified at the clinical site and eligibility was determined by each PI (74 US and International clinical sites).
Pre-assignment Details: Subjects who needed to washout omega-3 drugs/supplements or adjust or add a permitted statin, CAI or combination had an 8-week screening. All other subjects, including those on a stable statin, CAI or statin-CAI, or who needed to washout of bile acid sequestrants, fibrates, niacin and other lipid altering supplements had a 4-week screening period.
Groups:
- Olive Oil (Placebo Control): placebo : 4 capsules (1g) daily for 12 weeks
- Epanova 2 g: omefas : 2 capsules (1g) + 2 placebo daily for 12 weeks
- Epanova 3 g: omefas : 3 capsules (1g) + 1 placebo daily for 12 weeks
- Epanova 4 g: omefas : 4 capsules (1g)daily for 12 weeks
Period: Overall Study
Arm/Group | Olive Oil (Placebo Control) | Epanova 2 g | Epanova 3 g | Epanova 4 g
Started | 99 | 100 | 101 | 99
Completed | 94 | 93 | 87 | 90
Not Completed | 5 | 7 | 14 | 9

BASELINE CHARACTERISTICS:
Groups:
- Olive Oil (Placebo): placebo : 4 capsules (1g) daily for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Olive Oil (Placebo) | Epanova 2 g | Epanova 3 g | Epanova 4 g | Total
Number analyzed (Participants) | 99 | 100 | 101 | 99 | 399
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.8 (10.59) | 51.1 (9.79) | 51.2 (8.75) | 52.9 (10.92) | 51.5 (10.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 22 | 28 | 92
  Male | 77 | 80 | 79 | 71 | 307
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 4 | 7 | 25
  Not Hispanic or Latino | 93 | 92 | 97 | 92 | 374
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Fasting Serum Triglycerides
Description: The primary endpoints are the differences in mean percent changes from baseline to end-of-treatment in triglycerides between placebo and the 2g/day, 3g/day and 4g/day Epanova groups
Time Frame: 12 weeks
Population: The Intent-to-Treat (ITT) Population was comprised of all subjects who were randomized. In the event that randomized subjects terminated before treatment or had no post-treatment efficacy assessments, a modified ITT Population was implemented.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change from baseline
Arm/Group | Olive Oil (Placebo) | Epanova 2 g | Epanova 3 g | Epanova 4 g
Number analyzed (Participants) | 98 | 99 | 97 | 99
Percent change from baseline | -4.26 [-13.07 to 5.44] | -25.94 [-32.84 to -18.33] | -25.46 [-32.44 to -17.75] | -30.86 [-37.32 to -23.74]
Statistical Analysis 1: Comparison: Olive Oil (Placebo) vs Epanova 2 g; Test type: Superiority or Other; p = 0.005, ANCOVA p-value on ranked data — P-value adjusted with Dunnett's procedure for multiple comparisons of Epanova vs olive oil; ANCOVA model with baseline value as covariate, and treatment and user/non-user of lipid-altering drugs as factors; Placebo adjusted % change from baseline = -21.68, 95% CI 2-sided [-40.70 to -2.89] — ANCOVA on log-scale TG with baseline value as covariate and treatment and user/non-user of lipid-altering drugs as factors
Statistical Analysis 2: Comparison: Olive Oil (Placebo) vs Epanova 3 g; Test type: Superiority or Other; p = 0.007, ANCOVA p-value on ranked data — P-value adjusted with Dunnett's procedure for multiple comparisons of Epanova vs olive oil; ANCOVA model with baseline value as covariate, and treatment and user/non-user of lipid-altering drugs as factors; Placebo adjusted % change from baseline = -21.19, 95% CI 2-sided [-40.32 to -2.29] — ANCOVA on log-scale TG with baseline value as covariate, and treatment and user/non-user of lipid-altering drugs as factors
Statistical Analysis 3: Comparison: Olive Oil (Placebo) vs Epanova 4 g; Test type: Superiority or Other; p < 0.001, ANCOVA p-value on ranked data — P-value adjusted with Dunnett's procedure for multiple comparisons of Epanova vs olive oil; ANCOVA model with baseline value as covariate, and treatment and user/non-user of lipid-altering drugs as factors; Placebo adjusted % change from baseline = -26.60, 95% CI 2-sided [-45.12 to -8.38] — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Arm/Group | Olive Oil (Placebo) | Epanova 2 g | Epanova 3 g | Epanova 4 g
Serious Adverse Events (participants affected / at risk) | 2/99 | 1/100 | 4/101 | 0/99
Other Adverse Events (participants affected / at risk) | 5/99 | 23/100 | 18/101 | 16/99
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olive Oil (Placebo) (N=99) | Epanova 2 g (N=100) | Epanova 3 g (N=101) | Epanova 4 g (N=99)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Implantable defibrillator insertion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olive Oil (Placebo) (N=99) | Epanova 2 g (N=100) | Epanova 3 g (N=101) | Epanova 4 g (N=99)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 10 (12) | 6 (7) | 10 (11)
Nausea (Gastrointestinal disorders) | 1 (1) | 6 (9) | 9 (11) | 5 (5)
Nasopharyngitis (Infections and infestations) | 2 (3) | 7 (7) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Individual investigators may publish data arising from their own subjects. The PI will provide the Sponsor with copies of written publications (including abstracts and posters)at least 60 days in advance of submission. Data will be reviewed by all participating investigators prior to publication. The Sponsor will have 60 days to review all definitive publications, such as manuscripts and book chapters, and a minimum of 30 days to review all abstracts.